CLINICAL TRIAL: NCT03833011
Title: Postoperative Osteopathic Manipulative Treatment in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MediSys Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FHMCSURG01
Record Dates: First submitted 2019-01-18; First posted 2019-02-06 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Pain; Bariatric Surgery Candidate
MeSH Terms: conditions — Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no intervention (No Intervention)
- Osteopathic manipulation (Experimental)
  Interventions: Procedure: Osteopathic Manipulation

INTERVENTIONS:
Procedure: Osteopathic Manipulation — Osteopathic manipulation
  Arms: Osteopathic manipulation

SUMMARY:
Context Pain control is one of the most challenging problems encountered in postoperative period in bariatric patients. Currently there are no published studies evaluating Osteopathic Manipulative Treatment in bariatric surgery patients.

Objective The primary objective of this study is to determine whether Osteopathic Manipulative Treatment (OMT) can decrease pain score in bariatric patients. The secondary objective is whether OMT can improve patient satisfaction with overall treatment.

Design: A prospective randomized group controlled study.

Setting: A 293-bed non-for-profit teaching community hospital.

Methods Thirty-six patients scheduled for bariatric surgery as per ASMBS criteria were eligible for study from January 2017 through August 2018 at Flushing Hospital Medical Center, New York. Twelve patients were excluded.

Twenty-four patients were included into study and randomized to receive OMT(n=12) vs Control (n=12) intervention.

In Control group, patients received standard pain control protocol with morphine patient controlled analgesia pump (PCA) In OMT group, patients received standard postoperative pain protocol and OMT on postoperative day one. Three techniques were used (Sub-occipital Release, Thoracic Outlet Release, and Rib Raising). All patients received survey to complete prior to discharge measuring pain score (1-10), patient satisfaction score 1-4 (poor, fair, good, excellent) and data was analyzed.

ELIGIBILITY:
Inclusion criteria:

* Adults age 18 and older eligible for bariatric surgery as per American Society for Metabolic and Bariatric Surgery guidelines:
* BMI of at least 40, or greater than 100 pounds overweight.
* BMI of 35 or above and at least one or more obesity-related comorbidity such as type II diabetes, hypertension, sleep apnea and other respiratory disorders, non-alcoholic fatty liver disease, lipid abnormalities, gastrointestinal disorders, heart disease, or osteoarthritis.
* Inability to achieve a healthy weight loss sustained for a period of time with prior weight loss efforts.

Exclusion criteria:

* Age less than 18.
* Pregnant patients.
* Patients with history of chronic pain.
* Patients with diagnosed psychiatric disorders.
* Patients actively taking pain medication before surgery.
* Patients with prior surgical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in pain score | pre-intervention, post-op day 1, post-op day 2
  subjective measure of pain on a scale of 1-10

CONTACTS AND LOCATIONS:
Locations (1):
- Flushing Hospital, Flushing, New York, United States

IPD SHARING:
Plan to Share IPD: No